CLINICAL TRIAL: NCT04689646
Title: Mind Body Syndrome Therapy for the Treatment of Chronic Pain
Brief Title: Mind Body Syndrome Therapy for Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P000147
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain; Chronic Pain Syndrome
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Mind-Body Intervention 1, Mind-Body Intervention 2 and Usual Care
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) Participants will be partially blinded. Participants in the usual care arm will be blinded to the specifics of the interventions. Participants in Mind-Body Intervention 2 arm will be blinded to the specifics of the interventions. Intervention participants will be blinded to the specifics of the intervention until after they have been randomized into that arm. Data analysis will be conducted by persons who are completely blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mind-Body Intervention 1 (Experimental): Participants will receive a mind body educational based intervention to learn the techniques comprising intervention 1.
  Interventions: Behavioral: Mind Body Intervention 1
- Mind-Body Intervention 2 (Active Comparator): Participants will receive a mind body educational based intervention to learn the techniques comprising intervention 2.
  Interventions: Behavioral: Mind body intervention 2
- Usual Care (No Intervention): Participants will continue their usual care for 26 weeks

INTERVENTIONS:
Behavioral: Mind Body Intervention 1 — Mind body techniques for Intervention 1 will be taught in lectures and group discussion sessions.
  Arms: Mind-Body Intervention 1
Behavioral: Mind body intervention 2 — Mind body techniques for Intervention 2 will be taught in lectures and group and/or individual sessions.
  Arms: Mind-Body Intervention 2

SUMMARY:
The goal of this study is to determine if a mind-body intervention can help people suffering from chronic back pain. The study is a randomized, partially blinded trial examining the effectiveness of a mind body intervention in reducing disability from back pain and alleviating back pain in participants as compared to usual care and an active control (second mind body intervention). The investigators will secondarily investigate whether the intervention alleviates anxiety related to the pain and other quality of life parameters.

DETAILED DESCRIPTION:
The goal of this study is to determine if a mind-body intervention can help people suffering from chronic back pain. The study is a randomized, partially blinded trial examining the effectiveness of a mind body intervention in reducing disability from back pain and alleviating back pain in participants as compared to usual care (control arm) and an active control arm. The investigators will secondarily investigate whether the intervention alleviates anxiety related to the pain and other quality of life parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 ≥ years old
* Chronic back pain
* Pain persistent for a minimum of 3 days a week for the past three months prior to enrollment
* Willingness to consider mind-body intervention
* At least score of 2 or more on Roland Disability Questionnaire
* At least score of 3 or more back pain bothersomeness

Exclusion Criteria:

* Patients < 18 years of age
* Patients > 67 years of age
* Diagnosed organic disease as cause of pain, such as (but not limited) to malignancy, neurologic disorder (i.e., amyotrophic lateral sclerosis), cauda equina syndrome (note that pain related to disc disease is not an exclusion unless there are neurological impairments)
* Patients with a diagnosis of significant psychiatric co-morbidities such as schizophrenia, dementia, and bipolar disorder

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain Disability | 26 weeks
  Roland Morris Disability Index (Scale 0-24 with 24 being worst)

SECONDARY OUTCOMES:
Average pain | Baseline, 4, 8, 13, and 26 weeks after initiation of the study.
  Average pain as determined in the Brief Pain Inventory Survey (Scale 0-10 with 10 being worst)
Pain Bothersomeness (Back Specific): Brief Pain Inventory Survey | Baseline, 4 weeks, 8 weeks, 13 weeks, 26 weeks
  Back pain bothersomeness as determined from modified Brief Pain Inventory Survey. (Scale 0-10 with 10 being the worst
Pain bothersomeness: Brief Pain Inventory | Baseline, 4 weeks, 8 weeks, 13 weeks, 26 weeks
  Whole-body pain bothersomeness as determined from modified Brief Pain Inventory Survey (Scale of 0-10 with 10 being the worst)
Anxiety from pain | Baseline, 4 weeks, 8 weeks, 13 weeks, 26 weeks
  Anxiety from pain as determined from the Pain Anxiety Symptom Scale-20 survey (20 questions with scale of 0-5 with 5 being 'always' and 0 being 'never'
Self-reported hospital admissions | Baseline, 26 weeks
  Self reported. Number of pain-related hospital admissions, including emergency room visits
Complete resolution of pain disability | Baseline, 4 weeks, 8 weeks, 13 weeks, 26 weeks
  complete resolution of pain disability as measured by Roland Morris Disability (Scale 0-24 with 24 being worst)
Pain affecting enjoyment of life | Baseline, 4 weeks, 8 weeks, 13 weeks, 26 weeks
  Scale 0-10 with 10 being worst from Brief Pain Inventory
Complete resolution of back pain | Baseline, 4 weeks, 8 weeks, 13 weeks, 26 weeks
  complete resolution of pain as measured on scale 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No